CLINICAL TRIAL: NCT03402997
Title: Minimally Invasive Procedure for the Discrimination of Tissue Resistivity in Breast Cancer Patients
Brief Title: Tissue Resistivity in Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Ente Ospedaliero Cantonale, Bellinzona (Other)
Collaborators: Politecnico di Milano (Other); Clinical Trial Unit Ente Ospedaliero Cantonale (Other)
Responsible Party: Sponsor
Other Study IDs: OBV-GASTRO-001
Record Dates: First submitted 2018-01-11; First posted 2018-01-18 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Resistivity measurements: The resistivity measurements will be done by introducing the needle-probe into fresh healthy, peritumoral, and tumoral ex vivo tissues
  Interventions: Diagnostic Test: Resistivity measurement

INTERVENTIONS:
Diagnostic Test: Resistivity measurement — To measure and compare the tissue impedance values obtained by analysing ex vivo non-neoplastic (healthy and peritumoral) and neoplastic breast tissues

SUMMARY:
The resistivity measurements will be done by introducing a needle-probe into fresh healthy, peritumoral, and tumoral ex vivo tissues.

DETAILED DESCRIPTION:
Patients affected by breast cancer will have their tissue analysed immediately following their surgical excision for the treatment of breast cancer. Two probes will be used: a linear probe of 4 needle-electrodes positioned in a row that is able to perform Electrical Impedance Spectroscopy (EIS) measurements and a circular probe of 8 needle-electrodes arranged into a circular pattern that is able to generate cross sectional images (Electrical Impedance Tomography maps). Firstly, the linear probe will be inserted in the tumor parenchyma at a penetration depth of about 2 mm and the tissue impedance measurement will be performed along a broad spectrum of frequencies for few minutes. Approximately 10 seconds for each measurement will be needed. Subsequently, if the size of the tissue will allow it, the circular probe will be inserted in the tumor parenchyma at the same penetration depth and 10 cross sectional maps will be generated (approximately 30 seconds in total). Both information obtained using the linear and the circular probes will be integrated for a full characterization of the tissue under examination.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* First radiological diagnosis of breast adenocarcinoma needing a histological confirmation
* Written Informed Consent

Exclusion Criteria:

* Tumor mass diameter < 1 cm
* Surgical specimen (harbouring tumoral + peritumoral tissue) diameter < 2 cm

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: The target population of this study are female patients with first radiological diagnosis of breast cancer needing for surgery and subsequent histological examination to confirm the diagnosis.
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
Breat tissue characterization | 30 minutes from surgery
  Use of Electrical Impedance Spectroscopyuse (EIS) to characterize ex vivo non-neoplastic (healthy and peritumoral) and neoplastic breast tissues

SECONDARY OUTCOMES:
Evaluation of the precision of each EIS measurement | 30 minutes from surgery
  To evaluate the precision of each EIS measurement (healthy, peritumoral, cancerous) performed by the tissue impedance analyser in the same subject
Correlation between electrical and biological results | 30 minutes from surgery
  To correlate the electrical behaviour of the breast cancer tissue to pathological and biological information

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Regionale di Mendrisio, Mendrisio, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided